CLINICAL TRIAL: NCT02621086
Title: A Pilot Study to Assess the Tolerability of a Single, Ascending Dose of a Non-digestible Carbohydrate in Healthy Volunteers
Brief Title: Cellodextrin Tolerability Study
Acronym: CELLDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Dr, University of Nottingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RA3624; BB/L025019/1 (Other Grant/Funding Number: BBSRC)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: Oligosaccharide, Tolerability,
MeSH Terms: conditions — Obesity | interventions — cellodextrin

STUDY DESIGN:
Intervention Model Description: Ascending dose tolerability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Level 1 (Experimental): 10g of Cellodextrin
  Interventions: Dietary Supplement: Cellodextrin
- Level 2 (Experimental): 20g of Cellodextrin
  Interventions: Dietary Supplement: Cellodextrin
- Level 3 (Experimental): 30g of Cellodextrin
  Interventions: Dietary Supplement: Cellodextrin
- Level 4 (Experimental): 50g of Cellodextrin
  Interventions: Dietary Supplement: Cellodextrin

INTERVENTIONS:
Dietary Supplement: Cellodextrin — Gastrointestinal tolerability of single ascending doses of Cellodextrins

SUMMARY:
This is an initial pilot study to assess and investigate if any adverse symptoms occur (and also the severity of any symptoms) after consuming a food-grade Cellodextrin preparation. Volunteers will attend a short (around 30mins) medical screening visit, to make sure they are suitable to take part in the study. They will then attend 4 study visits (separated by at least a week) for around 9.5 hours each time. During the study visits 10, 20, 30, or 50g of Cellodextrin will be given as a single oral dose, in a milkshake drink, and any symptoms experienced will then be monitored via questionnaires during the study day and for the next 60 hrs, dietary intake will also be measured over this time.

DETAILED DESCRIPTION:
Cellodextrins are small-chain, non-absorbable, oligosaccharides that are produced from the incomplete hydrolysis of insoluble cellulose. Like other oligosaccharides they escape digestion in the small intestine as the human gut lacks the enzymes required to hydrolyse the β-links formed among the units of monosaccharides. However, Bifidobacterium in the caeco-colon possess the enzymes β-fructosidase and β-galactosidase which are needed to breakdown the carbohydrate chains to their constituent sugars, this serves the bacteria by providing energy for proliferation and also produces gases (Hydrogen, Carbon dioxide, and Methane, which are metabolically useless to the host), and short chain fatty acids (SCFA). This breakdown supplies an available energy estimated to be 1.5-2kcal/g, in comparison digestible carbohydrate produces 4kcal/g of available energy.

The prevalence of overweight and obesity is an increasing issue in the developed world and reduction of energy intake remains at the heart of the main treatments for obesity. Due to this there is an interest in identifying food ingredients that will combat dietary overconsumption. By replacing some of the digestible carbohydrates with non-digestible oligosaccharides it could be possible to reduce the caloric load of food by approximately 2kcal/g of carbohydrate, but still keep the taste and 'mouth-feel' of these reduced calorie products. Further benefits of the use of non-digestible oligosaccharides against dietary overconsumption include the contribution that these compounds could have on reducing appetite and voluntary food intake, which could further improve energy intake regulation. Oligosaccharides may increase satiety by bulking, by slowing gastric emptying, or by increasing production of Peptide-yy (PYY) and Glucagon like peptide-1 (GLP-1). The latter has been demonstrated in-vitro, where butyrate, one of the SCFA's produced in oligosaccharide break-down, increased PYY and Proglucagon production in rat epithelial cells. Little work has been done on the potential oligosaccharide effects on appetite. and assessment of the appetite effects and energy regulation potential of Cellodextrin in humans is even more limited. However, before studies to investigate this can be carried out, it is important to assess any gastro-intestinal disturbances that may occur at the doses which would be required.

The recommendation for total fibre intake is 18g/day in the United Kingdom (UK) although the actual UK average intake is lower than this, at an average of 13-15g/day. It is not known what the average daily oligosaccharide intake is in the UK, or whether the oligosaccharides are included in the total fibre estimates. However, because they are not digested within the small intestine, they can have a laxative effect, increasing the ease and/or frequency of laxation and excess intakes may cause diarrhoea and other gastrointestinal symptoms such as flatulence, bloating and abdominal discomfort. Intolerance symptoms can be due to the osmotic effect and/or fermentation; the osmotic effect may cause abdominal pain and eventually diarrhoea if the capacity of the colon to absorb water is exceeded. Moreover, fermentation produces gases that may also induce abdominal pain, bloating and excessive flatus. The tolerance of non-digestible oligosaccharides is usually very good, although the tolerance threshold depends on the type of oligosaccharide, the timing of consumption (e.g. after fasting or after a meal) and also individual factors such as absorption capacities, motility patterns, colonic responses and intestinal sensitivity. Polydextrose has been found to be tolerated at doses of 50g/day, resistant starch has a similar tolerability at acceptable doses of 45g/day, whereas galacto-oligosaccharide consumption of over 20g/day and fructo-oligosaccharide consumption of over 40g/day have been reported to cause diarrhoea.

The aim is to investigate initially whether Cellodextrin induces gastrointestinal symptoms in a UK cohort of healthy men and women and to what extent. This information can then be used to inform future volunteers as to the relative risks of developing these gastrointestinal problems and the severity of symptoms experienced. A descriptive pilot study will be carried out. Twelve healthy individuals (6 males and 6 females, 18-40y, with a BMI between 18 and 30kg/m2) will be recruited. Interested individuals will contact the investigators and be sent a copy of the information sheet before attending a medical screening. At the medical screening a full explanation of the study will be given and informed consent gained. A medical screening questionnaire will be administered, blood pressure measurements made and a 10ml blood sample will be taken via venepuncture by suitably qualified staff (analysed for full blood count, urea and electrolytes). If suitable, participants will attend the laboratory for up to 4 visits and to provide a fecal sample (for microbiota assessment) prior to attending the first study visit. Participants will arrive at the laboratory around 8am, fasted from midnight the night before, and will then complete a series of appetite and gastro-intestinal symptom questionnaires. They will be asked to empty their bladder and a 24hr urine collection will be started. After resting on a hospital bed for 15 min, a cannula will be sited for blood sampling. The participant will then consume 10, 20, 30 or 50g of Cellodextrin in a milkshake drink. They will repeat the questionnaires every 30 minutes for 180 minutes with 1ml of blood taken from the cannula every 15 minutes over this time. The cannula will then be removed and a standard snack given to stimulate gut motility and questionnaires (as before) will be completed after 210 and 240 minutes. A low fiber sandwich lunch will be provided at 240mins,and during the following 2 hours, questionnaires will be administered every 30 minutes and then again at 420 and 480mins. Participants will be given a diet and symptom diary to complete over the rest of the day and the following 48hrs after each study visit. Feedback forms will be administered if a participant withdraws from or completes the study. Further fecal samples will be collected between 24 and 48hrs after consumption of the 30g and 50g dose.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* BMI 18-30 kg/m2
* Healthy
* Random Blood Glucose concentration below 7.8mmol/l
* Ability to give written informed consent
* English speaking

Exclusion Criteria:

* Age <18 or >40 years
* Any significant medical condition
* Random Blood Glucose concentration above 7.8mmol/l
* Use of regular medication (other than oral contraceptive pill)
* Use of herbal supplements
* History of Irritable Bowel Syndrome (IBS), food intolerances or any gastrointestinal disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal discomfort | 60 hours
  Gastrointestinal discomfort assessed by visual analogue scale up to 60 hours post consumption of cellodextrin

SECONDARY OUTCOMES:
Diarrhoea | 60 Hours
  Bristol Stool Score used to assess change in bowel habit up to 60 hours after cellodextrin consumption
Subjective Appetite | 60 Hours
  Subjective appetite assessed periodically up to 60 hours after cellodextrin consumption using visual analogue scales
Energy Intake | 60 Hours
  Dietary energy intake assessed by diet diaries
Change in whole blood glucose concentration | 180 mins
  blood glucose response to the milkshake drink
Fecal microbiota | prior to exposure to the cellodextrin preparation
  assessment of the bacterial population in fecal samples
fecal microbiota | 48hrs
  change in bacterial population as a result of exposure to cellodextrins
Fluid balance | 24hrs
  fluid balance assessment for 24hrs after cellodextrin consumption

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — The University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No